CLINICAL TRIAL: NCT00397423
Title: Granulocyte-Colony Stimulating Factor Treatment for Amyotrophic Lateral Sclerosis: A Randomized Control Trial Study Assessing Clinical Response
Brief Title: G-CSF Treatment for Amyotrophic Lateral Sclerosis: A RCT Study Assessing Clinical Response
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R01-123456-1
Record Dates: First submitted 2006-11-08; First posted 2006-11-09 (Estimated); Last update posted 2007-11-28 (Estimated); Status verified 2007-11

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic Lateral Sclerosis; Granulocyte Colony Stimulating Factor; Randomized Control Trial Study
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor

ARMS (2):
- 1 (Active Comparator): 1,G-CSF,intervention
  Interventions: Drug: Granulocyte Colony Stimulating Factor
- 2 (Placebo Comparator): 2,NS,intervention
  Interventions: Drug: NS

INTERVENTIONS:
Drug: Granulocyte Colony Stimulating Factor — Granulocyte Colony Stimulating Factor,5ug/kg/day iH Qd*5 days,3 months interval for 4 times
  Arms: 1
Drug: NS — NS 1ml iH Qd*5 days, 3 months interval for 4 times
  Arms: 2

SUMMARY:
This study will examine the effectiveness of G-CSF in treating patients with amyotrophic lateral sclerosis (ALS) - a fatal neurological degenerative disease that causes adult-onset, progressive motor neurons loss in the spinal cord, brain stem and motor cortex. Patients develop progressive wasting and weakness of both upper and lower limbs, bulbar and respiratory muscles. Usually death from respiratory failure typically is within 3-5 years of diagnosis. Although there are various treatments for ALS, riluzole is the only approved treatment to delay the disease progression. G-CSF is an approved drug that is used to increase white blood cell counts. Moreover, G-CSF and its receptor are expressed by neurons. It acts anti-apoptosis by activating several protective pathways, stimulates neuronal differentiation of adult neural stem cells in the brain, and improves long-term recovery. G-CSF is a novel neurotrophic factor, and a highly attractive candidate for the treatment of neurodegenerative conditions such as ALS.

Patients 18 to 65 years of age who have had mild to moderately severe ALS for 0.5 to 2 years of duration may be eligible for this study. Candidates will be screened with a medical history and possible review of medical records, physical examination, blood test, urine and stool analyses, electrocardiogram, electrophysiological examination, neurological imaging and, for women, a pregnancy test.

Participants will have drug therapy according to randomized number. One group receives G-CSF while other group receives placebo. All of the participants receive riluzole treatment. For the procedure, patients are given a medication to lessen anxiety and any discomfort. Patients receive drug injections every 3 months for 5 days. The G-CSF dosage is 5μg/kg/day. Physical examination and interview, Appel ALS scale and ALS-Functional Rating Scale will be done in 14, 28 days and 3, 6, 9, 12 months. Electrophysiological examination will be tested per 3 months. Blood samples will be collected on treat 5, 14, 28 days and 3, 6, 9, 12 months.

ELIGIBILITY:
Inclusion Criteria:

* All subjects must have a verifiable diagnosis of ALS of 0.5 to 2 years' duration. The diagnosis must be supported by the Revised Criteria of the World Federation of Neurology. The grades of diagnosis must be clinically definite ALS or clinically probable ALS.
* All subjects must be over age 18 and below 65.
* The ALS is mildly to moderate based on ALS Health State Scale.
* Electrophysiological features show CMAP amplitude of motor nerve normal or mild declining.
* Serum creatine kinase is normal or mild upper, less than 500U/L.

Exclusion Criteria:

* If anyone of the above eligibility requirements is not met
* Use of any other investigational agent within 30 days beginning the treatment phase of this study
* Severe cardiac, pulmonary, hepatic or/and hematic disease
* HIV positivity or signs and symptoms consistent with HIV infection
* Pregnant or nursing women
* History of cancer with less than 5 years documentation of a disease-free state
* History of anaphylactic reaction or hypersensitivity to G-CSF or proteins derived from E.coli
* Alcohol or drug abuse in recent 1 year
* Can't understand or obey the rules of treatment
* Blood donor in recent 30 days

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-12; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
the mean rate of decline of ALS-FRS score | 12 months

SECONDARY OUTCOMES:
the mean rate decline of the AARS score | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Dongsheng Fan, MD, Study Chair — Peking University Third Hospital
Locations (1):
- Dongsheng Fan, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Fan DS, Zhang J, Deng M, Kang DX, Zheng JY, Xu YS, Lu M, Fu Y, Shen Y, Zhang YS, Zhang HG. [Basic and clinical researches on amyotrophic lateral sclerosis/motor neuron disease]. Beijing Da Xue Xue Bao Yi Xue Ban. 2009 Jun 18;41(3):279-81. Chinese. PMID 19727208